CLINICAL TRIAL: NCT01662323
Title: Therapy OPtimization Heart Failure Utrecht
Brief Title: Study to Improve the Treatment of Patients With Heart Failure by General Practitioners
Acronym: TOPHU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Julius Center (Other)
Collaborators: Agis Zorgverzekeringen (Other)
Responsible Party: Principal Investigator, Drs. Mark M J Valk, assistant professor, Julius Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOPHU01
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Heart Failure
Keywords: Heart failure, general practitioner, medical therapy, quality of live
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training of the GP's, intervention (Active Comparator): General practitioners are trained to diagnose and treat heart failure according the recommendations of the NHG-standard.
  Interventions: Behavioral: GP's treating HF according the dutch guidelines
- Controle (Active Comparator): General practitioners giving care as usual to their heart failure patients.
  Interventions: Behavioral: GP's treating HF according the dutch guidelines

INTERVENTIONS:
Behavioral: GP's treating HF according the dutch guidelines

SUMMARY:
The purpose of this study is to determine whether it is possible to improve the care of general practitioners for patients with heart failure. The investigators try to reach that goal by training the GP's for 90 minutes in uptitrating the recommended medication according the guidelines. After 6 month the investigators ask the patients to fill out a questionary. The investigators ask them about their quality of live.

ELIGIBILITY:
Inclusion Criteria:

* Do have a general practitioners diagnosis heart failure mentioned twice in the electronical medical file.

Exclusion Criteria:

* Incapacitated patients with a life expectancy of less than 2 months
* Seniles
* Patients who do not speak the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
proportion recommended medication for patients with heart failure | up to 6 months
  the proportion patient who got at the end of the study the tree medicaments which should be prescribed to a patient with heart failure.

SECONDARY OUTCOMES:
QoL | up to 1 year
  Measurement of quality of live six months after uptitration of the recommended medication.

REFERENCES:
- [Derived] Valk MJ, Hoes AW, Mosterd A, Landman MA, Broekhuizen BD, Rutten FH. Rationale, design and baseline results of the Treatment Optimisation in Primary care of Heart failure in the Utrecht region (TOPHU) study: a cluster randomised controlled trial. BMC Fam Pract. 2015 Oct 7;16:130. doi: 10.1186/s12875-015-0347-1. PMID 26446696
- [Derived] Valk MJ, Broekhuizen BD, Mosterd A, Zuithoff NP, Hoes AW, Rutten FH. COPD in patients with stable heart failure in the primary care setting. Int J Chron Obstruct Pulmon Dis. 2015 Jun 26;10:1219-24. doi: 10.2147/COPD.S77085. eCollection 2015. PMID 26170650